CLINICAL TRIAL: NCT01000688
Title: The Effect of Vildagliptin on Endothelium-dependent Vasodilatation. A Double Blind Cross-over Study in Type 2 Diabetes Mellitus.
Brief Title: Vildagliptin and Endothelium-dependent Vasodilatation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Prof. Dr. C.J. Tack, UMC St Radboud
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: VILD1
Record Dates: First submitted 2009-10-21; First posted 2009-10-23 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2009-10

CONDITIONS: Type 2 Diabetes; Endothelial Dysfunction
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; Acarbose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vildagliptin treatment first, acarbose treatment second (Experimental)
  Interventions: Drug: vildagliptin + acarbose
- acarbose treatment first, vildagliptin treatment second (Experimental)
  Interventions: Drug: acarbose + vildagliptin

INTERVENTIONS:
Drug: vildagliptin + acarbose — 4 week treatment
  Arms: vildagliptin treatment first, acarbose treatment second
Drug: acarbose + vildagliptin — 4 week treatment
  Arms: acarbose treatment first, vildagliptin treatment second

SUMMARY:
Rationale: Cardiovascular complications in type 2 diabetes are the leading cause of morbidity and mortality associated with the disease. Endothelial dysfunction is regarded as an important factor in these vascular complications.

The introduction of glucagon-like peptide-1 (GLP-1) analogues and dipeptidyl peptidase IV (DPP-IV) inhibitors for the treatment of type 2 diabetes is of special interest because of possible influences on endothelial function. Numerous reports have shown that GLP-1 improves endothelial function.

Objective: To determine whether a four week treatment with vildagliptin compared to acarbose improves endothelial dysfunction in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Age 35-75 years
* Treatment with metformin monotherapy or metformin combination therapy
* HbA1c <8.0%

Exclusion Criteria:

* Renal disease defined as creatinine level > 130 umol/l
* Liver disease defined as aspartate aminotransferase or alanine aminotransferase level of more than three times the upper limit of normal range
* Current use of acetylsalicylic acid or vitamine K antagonists
* History of smoking within the past year
* History of or current abuse of drugs or alcohol
* History of heartfailure (NYHA class III or IV)
* Abnormalities on ECG that might interfere with current study protocol
* Pregnancy or breastfeeding
* Inability to understand the nature and extent of the trial and procedures required
* Presence of any medical condition that might interfere with the current study protocol
* Participation in a drug trial within 60 days prior to the first dose

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Forearm vasodilator response to intra-arterial infusion of acetylcholine (endothelium-dependent) following treatment with vildagliptin and following active control with acarbose | 8 weeks

SECONDARY OUTCOMES:
Effect of vildagliptin on inflammatory markers and adipokines | 8 weeks
Effect of vildagliptin on fat cell morphology and gene expression | 8 weeks
Effect of vildagliptin on ex vivo mononuclear cell responses to various stimuli | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: C.J. Tack, MD, PhD, Prof. of Diabetology, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] van Poppel PC, Gresnigt MS, Smits P, Netea MG, Tack CJ. The dipeptidyl peptidase-4 inhibitor vildagliptin does not affect ex vivo cytokine response and lymphocyte function in patients with type 2 diabetes mellitus. Diabetes Res Clin Pract. 2014 Mar;103(3):395-401. doi: 10.1016/j.diabres.2013.12.039. Epub 2014 Jan 3. PMID 24485397